CLINICAL TRIAL: NCT02072902
Title: Diabetes, Glucose Control, Glucose Lowering Medications, and Cancer Risk: A 10-year Population-based Historical Cohort
Acronym: DBCA
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Other Study IDs: SHEBA-14-0050-RD-CTIL
Record Dates: First submitted 2014-02-12; First posted 2014-02-27 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Cancer
Keywords: Cohort; Historical; Prospective; Medications; Observational; Glucose; Control
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 11 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- diabetes free: No intervention
- Diabetes prevalent: The exposure is diabetes morbidity present at study entery
- Diabetes incidence: The exposure is diabetes incidence during study follow up

SUMMARY:
This is a large nationwide population study, with 10 year follow-up, of the effect of diabetes, metabolic control and a large number of glucose-lowering medications, on total and site-specific cancer incidence and survival.

The study is based on electronic medical records from the largest Israeli health maintenance organization in Israel, Clalit Health Services. 2,301,990 insurees age 21 years old or above at study entry, January 2002 will be included. Four study groups will be established according to the prevalence of diabetes and/or cancer on that date: neither diabetes nor cancer; prevalent diabetes but not cancer; prevalent cancer but not diabetes; both diabetes and cancer prevalence. Subjects free of diabetes at study entry will be followed for diabetes incidence, and all four groups will be followed until December 2012 for study outcomes. The cohort data file will be linked to the Israel National Cancer Registry for cancer morbidity.

We will compare, after adjustment, all and site-specific cancer rates between individuals with and without diabetes; and investigate if metabolic control, as indicated by HbA1c and blood glucose levels, is related to cancer risk. Using time-dependent Cox proportionate hazard models, we will then evaluate differences in outcomes that associate with the use of one or a combination of glucose-lowering treatments, while stratifying by those who were already diagnosed with diabetes at study entry, and those diagnosed during follow-up. Data for a large number of potential confounding variables, including BMI, plasma glucose, HbA1c, hormone replacement therapy and comorbidities will help mitigate allocation bias. The accessibility and uniformity of the healthcare provided by Clalit Health Services, as well as data on cancer screening tests, will minimize the risk of surveillance bias.

DETAILED DESCRIPTION:
The study was based on electronic records from the largest health maintenance organization in Israel, Clalit Health Services, which insures and provides healthcare to 55% (3.9 million) of the nation's population. All persons between 21 and 90 years and registered with Clalit on January 1, 2002 (the date of study entry), without a previous history of cancer, were included in a closed cohort that was followed until December 31 2012.

All individuals were followed for cancer incidence, which was ascertained by record linkage to the Israel National Cancer Registry, established in 1960. The registry has benefited since 1982 from a national law mandating registration of cancer, and has greater than 95% coverage of solid tumors, and approximately 85% coverage of hematologic cancers [34].

Definitions of diabetes: Incident diabetes was defined as fulfillment of at least one of the following six criteria during 2002-12: (1) diabetes recorded in the Clalit Chronic Disease Registry; (2) a physician's diagnosis of diabetes, and one plasma glucose test > 125 mg/dL within 12 months; (3) one HbA1c measurement > 6.5%; (4) 2-hour plasma glucose level during an oral glucose tolerance test ≥ 200 mg/dL; (5) 3 or more purchases of glucose-lowering medication within 12 months; (6) 2 plasma glucose measurements > 125 mg/dL within 12 months. The date of the earliest defining criterion was considered the date of diagnosis.

Prevalent diabetes was defined as being recorded with diabetes in the Clalit Chronic Disease Registry on study entry, or fulfilling criterion #5 above (information on medication use was available from 1998) before study entry.

Types of cancer: The following cancers were investigated: liver (ICD-O-3 codes C22.0 and C22.1), pancreas (C25.0-C25.9), gallbladder (C23.9-C24.9), endometrium (C54.0-C54.9, C55.9), stomach (C16.0-C16.9), kidney (C64.9, C65.9, C66.9., C68.0-C68.9), benign brain and central nervous system (C70.0-C72.9 with behavior code 0), malignant brain (C70.0-C72.9 with behavior code 3), multiple myeloma (C42.1 with relevant morphology codes), colorectum (C18.0-C21.8), non-Hodgkin lymphoma (C02.4, C09.8. C09.9, C11.1, C14.2, C37.9, C42.2, C77 and all other sites for extra-nodal Non Hodgkin's lymphoma), lung (all: C34.0-C34.9), adenocarcinoma, squamous cell), leukemia (C42.0, C42.1, C42.2 with relevant morphology codes), ovary (C56.9), bladder (C67.0-C67.9), breast (C50.0-C50.9), thyroid (C73.9) and prostate (C61.9). Apart from benign brain tumors, all cancers included in the analysis were coded as invasive (behavior code = 3).

ELIGIBILITY:
Inclusion Criteria:

* Aged older than 21 and younger than 90 at study entry, January 1, 2002
* Insured by Clalit Health Services

Exclusion Criteria:

* Under age 21 at January 1, 2002
* Over age 90 at January 1, 2002

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will include all individuals who were aged 21 years or older at study entry, January 1, 2002, and who were insured by Clalit Health Services, from one year prior to study entry, until the end of the study period, December 31, 2012, or until death, for those who did not survive until the end of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 2188669 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hazard ratios for all-site and site specific cancer | The population will be followed historically for incidence of cancer for a period of up to 11 years.
  The population will be followed historically for a period of up to 11 years whichever came first, cancer incidence, mortality, age 90, or end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Dankner, MD MPH, Principal Investigator — Gertner Institute, Sheba Medical Center
Locations (1):
- The Gertner Institute for Epidemiology and Health Policy Research, Ramat Gan, Israel

REFERENCES:
- [Background] Dankner R, Balicer R, Boffetta P, Boker LK, Wallenstein S, Freedman L, Goldfracht M, Roth J, Tamler R, LeRoith D. Diabetes, glucose control, glucose lowering medications, and cancer risk: a 10-year population-based historical cohort. BMC Cancer. 2012 Aug 23;12:364. doi: 10.1186/1471-2407-12-364. PMID 22917080
- [Result] Dankner R, Boffetta P, Keinan-Boker L, Balicer RD, Berlin A, Olmer L, Murad H, Silverman B, Hoshen M, Freedman LS. Diabetes, prostate cancer screening and risk of low- and high-grade prostate cancer: an 11 year historical population follow-up study of more than 1 million men. Diabetologia. 2016 Aug;59(8):1683-91. doi: 10.1007/s00125-016-3972-x. Epub 2016 May 17. PMID 27189066
- [Result] Dankner R, Boffetta P, Balicer RD, Boker LK, Sadeh M, Berlin A, Olmer L, Goldfracht M, Freedman LS. Time-Dependent Risk of Cancer After a Diabetes Diagnosis in a Cohort of 2.3 Million Adults. Am J Epidemiol. 2016 Jun 15;183(12):1098-106. doi: 10.1093/aje/kwv290. Epub 2016 Jun 2. PMID 27257115
- [Derived] Dankner R, Murad H, Agay N, Olmer L, Freedman LS. Glucagon-Like Peptide-1 Receptor Agonists and Pancreatic Cancer Risk in Patients With Type 2 Diabetes. JAMA Netw Open. 2024 Jan 2;7(1):e2350408. doi: 10.1001/jamanetworkopen.2023.50408. PMID 38175642
- [Derived] Dankner R, Freedman LS, Gerstein HC, Roth J, Keinan-Boker L. Newly diagnosed type 2 diabetes may serve as a potential marker for pancreatic cancer. Diabetes Metab Res Rev. 2018 Sep;34(6):e3018. doi: 10.1002/dmrr.3018. Epub 2018 Jun 17. PMID 29673046